CLINICAL TRIAL: NCT06961175
Title: Observational Study of Preoperative or Extracorporeal Circulation-induced Platelet Dysfunction Assessed by Thromboelastography in Non-antiplatelet-treated Patients Undergoing Cardiovascular Surgery (DISPLATEG Study)
Brief Title: Observational Study of Platelet Dysfunction Assessed by Thromboelastography in Cardiovascular Surgery (DISPLATEG)
Acronym: DISPLATEG
Status: Recruiting | Type: Observational
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Responsible Party: Principal Investigator, Jose Alfonso Sastre, Principal Investigator, Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León
Other Study IDs: PI 2025 03 1850
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Blood Platelet Disorders; Cardiac Surgery; Postoperative Bleeding
MeSH Terms: conditions — Blood Platelet Disorders; Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perioperative bleeding requiring blood transfusion is common during cardiovascular surgery, especially in procedures requiring cardiopulmonary bypass. Adenosine diphosphate (ADP) plays a fundamental role in platelet function. Several studies have shown that some patients not receiving antiplatelet therapy undergoing cardiovascular surgery have decreased platelet ADP receptor activity; the prevalence of this condition can be as high as 36%.

Furthermore, extracorporeal circulation itself has been shown to cause a reduction in platelet function. Platelet dysfunction due to reduced platelet receptor activity after cardiac surgery is potentially a common cause of bleeding, perioperative blood transfusion, and surgical reexploration in patients not receiving antiplatelet agents. However, these studies are conducted with few patients and present some contradictory results, so the evidence is still scarce.

The study hypothesis is that preoperative platelet dysfunction for ADP measured by TEG® Platelet Mapping™ is associated with a higher incidence of moderate-severe bleeding after CPB in patients undergoing cardiovascular surgery.

DETAILED DESCRIPTION:
Perioperative bleeding requiring blood transfusion is common during cardiovascular surgery, especially in procedures requiring cardiopulmonary bypass. Cardiac surgery is one of the groups that uses the most blood products, with 20% to 40% of patients requiring transfusions for routine procedures. Various publications have shown that these types of procedures consume between 10% and 15% of the blood supply in Western countries.

The etiology of bleeding and coagulopathy is generally multifactorial and may result from hemodilution, surgical losses, residual effects of anticoagulant and antiplatelet drugs, activation of tissue factor in the extrinsic system, contact activation of the intrinsic system in components of the extracorporeal circulation (ECC) circuit, and the presence of residual heparin after CPB. This process can lead to hyperfibrinolysis, reduced platelet count and function, decreased fibrinogen concentration, and depletion of coagulation factors, culminating in impaired thrombin generation. Surgical trauma and the CPB circuit itself produce an increase in inflammatory cytokines, interleukins, and tumor necrosis factor, which in turn contribute to increased release and activation of coagulation factors, as well as dysregulated fibrinolysis.

Adenosine diphosphate (ADP) plays a fundamental role in platelet function. When secreted from the platelet-dense granules where it is stored, it amplifies platelet responses induced by other platelet agonists and stabilizes platelet aggregates. Several studies have shown that some patients not receiving antiplatelet therapy undergoing cardiovascular surgery have decreased platelet ADP receptor activity; the prevalence of this condition can be as high as 36%. In healthy blood donors, an average reduction in this activity of 18% has been shown, as measured by TEG® Platelet Mapping™ (Haemoscope Corporation, Niles, Illinois, USA) (0-58%). Furthermore, extracorporeal circulation itself has been shown to cause a reduction in platelet function, as measured by both the TEG® Platelet Mapping™ technique and aggregometry (Multiplate®). Platelet dysfunction due to reduced platelet receptor activity after cardiac surgery is potentially a common cause of bleeding, perioperative blood transfusion, and surgical reexploration in both patients not receiving antiplatelet agents and those treated with clopidogrel. However, these studies were conducted with small numbers of patients and presented some contradictory results, so the evidence is still scarce.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Patients undergoing elective surgery under CPB.
* Patients must be duly informed and have signed the informed consent form.
* ASA status I-IV.
* Sufficient intellectual capacity to understand the procedure.
* Normal preoperative coagulation study and platelet count.

Exclusion Criteria:

* Failure to meet the criteria listed above.
* Preoperative administration of antiplatelet agents with an inadequate washout period (5 days for clopidogrel and ticagrelor and 7 days for plasugrel).
* Preoperative administration of anticoagulants with an inadequate washout period.
* Thrombopenia <100,000 platelets or anemia <11 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population undergoing scheduled for cardiovascular surgery at the University Hospital of Salamanca will be taken as the reference population.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Amount of postoperative bleeding | 24 hours
  Amount of blood collected in drains after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: José A. Sastre, Study Director — Salamanca University Hospital
Locations (1):
- Salamanca University Hospital, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No